CLINICAL TRIAL: NCT03344952
Title: Long Term Improvement on GMFCS Level of Patients With Cerebral Palsy Treated by an Integrated Approach of Repeated Botulinum Toxin-A Injections
Brief Title: Improvement on GMFCS Level of Patients With Cerebral Palsy Treated by Repeated Botulinum Toxin-A
Status: Completed | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Nigar Dursun, Professor, MD, Kocaeli University
Other Study IDs: KU GOKAEK 2017/90
Record Dates: First submitted 2017-11-14; First posted 2017-11-17 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA; Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

INTERVENTIONS:
Drug: Botulinum toxin type A — Repeated injections to hypertonic muscles
  Other Names: Botox, Dysport
Other: Physical therapy — 3 weeks intensive program 1 week -10 days after BoNT-A injections

SUMMARY:
The aim of this retrospective, monocenter, observational study is to evaluate the changes in GMFCS levels of children with cerebral palsy (CP) who received repeated Botulinum Toxin-A (BoNT-A) injections in the lower limb(s) with an integrated treatment approach in Kocaeli University Department of PMR and Izmit Rehabilitation Center.

DETAILED DESCRIPTION:
It is generally agreed that children with CP reach their gross motor potential by the age of 3.5-5 and a child or young person over the age of 5 years will not improve their GMFCS level. BoNT-A is an important treatment in children with CP because it is safe in young children and allows combined treatment. The reduction in muscle tone by this selective treatment provides an opportunity to allow and optimize the effects of other treatments including orthoses, casting, conventional therapies and activity based functional trainings. For this reason, BoNT-A injections are always combined with other therapies in Kocaeli University Department of PMR and Izmit Rehabilitation Center. Adjunctive treatments in this department consists of serial casting, orthotics, physical therapy, occupational therapy, cognitive rehabilitation, special educational programs, non invasive brain stimulation with transcranial direct current, neurofeedback, biofeedback, electrical stimulation and other physical therapy modalities, activity based models including functional ambulatory training, constraint induced therapy, bilateral therapy, hippotherapy, music therapy by singing or playing percussive instruments or moving and dancing to music, and robotic rehabilitation. Individualized intensive combined treatment plan was applied by an appropriate neurorehab team to each patient within the department as a half day or full day program usually for 3 weeks starting 1 week or 10 days after BONT-A injections. In thıs retrospective, monocenter, observational study a software database program will be developed and all the present data about the demographic and clinic properties of the patients, all information about BoNT-A injections including safety and applied adjunctive treatments will be entered and reviewed.

ELIGIBILITY:
Inclusion Criteria:

* All children with a diagnosis of cerebral palsy with respect to Rosenbaum criteria
* Children who received at least 2 repeated BoNT-A injections to lower limb(s) as well as an integrated treatment approach (an intensive therapy protocol consisted of a half day or entire day program in Kocaeli University Department of PMR and Izmit Rehabilitation Center) within the last 10 years

Exclusion Criteria:

* Children who did not receive repeated injections
* Children who did not receive an intensive therapy protocol

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children diagnosis of cerebral palsy with respect to Rosenbaum criteria having received at least 2 repeated BoNT-A injections to lower limb(s) as well as an integrated treatment approach (an intensive therapy protocol consisted of a half day or entire day program in Kocaeli University Department of PMR and Izmit Rehabilitation Center) within the last 10 years
Sampling Method: Non-Probability Sample
Enrollment: 503 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-11-09 (Actual)

PRIMARY OUTCOMES:
Gross Motor Functional Classification System (GMFCS) | 10 years
  Motor development

SECONDARY OUTCOMES:
Modified Ashworth Scale (MAS) | Before and 4-6 weeks after each injection
  Assessment of tone
Angle of catch (XV3) of Modified Tardieu Scale (MTS) | Before and 4-6 weeks after each injection
  Assessment of spasticity
Observational Gait Scale (OGS) | Before and 4-6 weeks after each injection
  OGS is a measurement tool for analysis of gait consisting of seven gait parameters with a total score of 20.

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No